CLINICAL TRIAL: NCT02158273
Title: Medication Development in Alcoholism: Investigating PPAR Agonists
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, PI, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AA012602-14A1; R01AA012602 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-06-06 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Alcoholism
Keywords: Alcohol; Relapse
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Sugars; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRICOR (fenofibrate) (Active Comparator)
  Interventions: Drug: TRICOR (fenofibrate)
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Sugar Pill — 145 mg/day, oral pill, 9 days
  Arms: Sugar Pill
Drug: TRICOR (fenofibrate) — 145 mg/day, oral pill, 9 days
  Other Names: Fenofibrate; Fenoglide; Trilipix; Lipofen
  Arms: TRICOR (fenofibrate)

SUMMARY:
The primary hypotheses under test are that alcohol dependent subjects treated with fenofibrate will report decreased craving for alcohol following cue-exposure in the laboratory and report less drinking post treatment relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, 18-65 years of age
* Meets DSM-V criteria for Alcohol Use Disorder ≥ moderate severity and DSM-IV criteria for current alcohol dependence
* Subjects will not be seeking treatment because the medication studies are not treatment trials
* Subjects must be abstinent a minimum of 3 days (but not more than 7 days) prior to the human lab session
* Negative BAC and a CIWA score of < 9 at screening and time of lab session to eliminate acute alcohol or withdrawal effects on dependent measures
* In acceptable health in the judgment of the study physician, on the basis of interview, medical history, physical exam, ECG, urine test and lab tests
* Females with childbearing potential must have a negative serum pregnancy test on the screening visit with a negative urine pregnancy test at randomization and agree to use an effective method of birth control for the study duration and two weeks thereafter.
* Subjects must be able to complete and understand questionnaires and study procedures in English and sign an informed consent
* Willingness to comply with the provisions of the protocol and take daily oral medication

Exclusion Criteria:

* Subjects with a medical condition that contraindicates the administration of fenofibrate or that will increase potential risk as determined by the Study Physician.
* GGT more than 3 times the upper limit of normal
* Female subjects with childbearing potential who are pregnant, nursing, or refuse to use an effective method of birth control for the duration of the study and two weeks thereafter
* Meets DSM-V criteria for a major Axis I disorder including mood or anxiety disorders or substance use disorders (e.g., cocaine, amphetamines, heroin, PCP) other than alcohol or nicotine
* Has a positive UDS at screening or Visit 3 (laboratory session)
* Treatment within the month prior to screening with an investigational drug, vaccine or drugs that may influence study outcomes, or drugs that may pose a safety risk as determined by the Study Physician.
* History of hypersensitivity to the study drugs or the ingredients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- Susan Quello, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenofibrate: TRICOR (fenofibrate): 145 mg/day, oral pill, 9 days
- Placebo: Matched Placebo
Period: Overall Study
Arm/Group | Fenofibrate | Placebo
Started | 25 | 25
Completed | 22 | 22
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenofibrate | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.52 (12.40) | 36.64 (11.84) | 37.58 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale of Craving to Drink at 1 Week Following Administration of Fenofibrate or Placebo During the Double-Blind Period
Description: The four Visual Analog Scale (VAS) questions assess domains of alcohol craving: the intention to drink, loss of control, relief craving, and urge intensity. Each VAS scale item score ranges from 1-20 where a one indicates no craving and 20 indicates severe craving; thus, a higher score indicates a worse outcome. Total is a summation of the four VAS item scores (i.e. Intent, Impulse, Relief, Strength) and ranges in value from 4-80 with higher scores indicative of a worse outcome.
Time Frame: 1 week following administration of fenofibrate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fenofibrate | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  Strength | 8.94 (5.69) | 10.37 (6.01)
  Intent | 9.83 (6.39) | 11.03 (6.24)
  Impulse | 6.87 (6.55) | 6.98 (5.62)
  Relief | 6.92 (6.43) | 8.86 (6.00)
  Total | 32.56 (23.57) | 37.24 (21.84)

2. Secondary Outcome: Change From Baseline in Standard Drinks Per Week at 1 Week
Description: Standard drinks are equivalent to 14 grams of pure alcohol and number of drinks are assessed with Timeline Follow-Back (TLFB) methods. Change = (Week 1 - Baseline). More negative values indicate less use of alcohol.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: drinks/week
Arm/Group | Fenofibrate | Placebo
Number analyzed (Participants) | 22 | 22
drinks/week
  Drinks/week Baseline | 51.21 (27.24) | 47.22 (16.55)
  Drinks/week Week 1 | 31.77 (19.53) | 28.24 (11.44)
  Drinks/week Change | -19.44 (19.16) | -18.98 (12.07)

ADVERSE EVENTS:
Arm/Group | Fenofibrate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fenofibrate (N=25) | Placebo (N=25)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No